CLINICAL TRIAL: NCT03198442
Title: Role of Dedicated Breast PET in the Characterisation of Indeterminate Breast Lesions on MRI Requiring a Second-look Ultrasound - a Feasibility Study
Brief Title: Breast PET Feasibility
Acronym: Breast PET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 9702 Breast PET Feasibility; 16/LO/0507 (Other: NHS Health Research Authority)
Record Dates: First submitted 2017-03-16; First posted 2017-06-26 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Breast Neoplasm Female

STUDY DESIGN:
Intervention Model Description: Small cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast PET (Experimental): PET imaging of breast with patient in prone position.
  Interventions: Procedure: F-18 FDG breast PET scan

INTERVENTIONS:
Procedure: F-18 FDG breast PET scan
  Other Names: MAMMI

SUMMARY:
Breast PET may be able to help in the diagnostic pathway in patients to determine which ones need to go on to have a second look ultrasound +/- biopsy and those who need to be sent for MRI guided biopsy. This may reduce the need to create more anxiety and uncertainty in this group of patients, already extremely stressed by the recent diagnosis of breast cancer.This study involves a single trial visit the Royal Free Hospital for imaging. Participants will need to lie flat for up to 30 minutes on the PET-CT camera and up to 30 minutes on the MAMMI. They will be advised not to take part in this study if they are unable to lie flat on their back and their front for this length of time or if they are claustrophobic. They will be offered the opportunity to see the PET-CT scanner and the MAMMI before deciding to consent to the trial.

DETAILED DESCRIPTION:
This study involves a single trial visit the Royal Free Hospital for imaging. Participants will need to lie flat for up to 30 minutes on the PET-CT camera and up to 30 minutes on the MAMMI. They will be advised not to take part in this study if they are unable to lie flat on their back and their front for this length of time or if they are claustrophobic. They will be offered the opportunity to see the PET-CT scanner and the MAMMI before deciding to consent to the trial.

Participants will be exposed to a radiation dose from the radioactive tracer F-18 FDG that is injected into the vein before the scan and from the CT exposures during the scan. The dose associated with the injection of about 3 MBq/kg of F-18 FDG is in the range of 4-7mSv. A CT will be performed over the thorax to allow attenuation correction of PET images and localisation of tracer uptake. The dose from the thorax CT will be patient dependent but the mean dose to a patient undergoing this type of scan is 2.1mSv. A whole body CT will be performed from the base of the skull to mid-thigh to plan the bed positions for the whole body emission scan and to allow attenuation correction of PET images and localisation of tracer uptake. The dose from the whole body CT will be patient dependent but the mean dose to a patient undergoing this type of scan is 5.2mSv.The total radiation dose participants will be exposed to is in the range of 11.3-14.3mSv. This is equivalent to 4-5.3 years of background radiation to which individuals in the UK are regularly exposed. This would amount to an increased lifetime risk of cancer of approximately 1 in 1250 in a standard population. These risks are compared to a normal lifetime risk of cancer of 1 in 3.

The half-life of F-18 is 110 minutes. The duration of the scan will be up to 120 minutes post injection. The activity within the patient will have reduced by more than 50% through radioactive decay alone by the time they leave the department and will be further reduced by excretion in urine. As with standard clinical administration of F-18, patients will not need to follow any special restrictions once leaving the department.

The CT scanning protocols used in the trial PET-CT are the standard clinical protocols used in the nuclear medicine department and have been developed with a view to minimising the dose to the patient as far as possible. All women of childbearing potential will undergo a pregnancy test on the day of the scan before the injection of the radioactive tracer in order to rule out any risk to a potential foetus. Any woman of childbearing potential who is found to be pregnant or will not consent to a pregnancy test will be excluded from the trial.

Very rarely, individuals may develop an allergic reaction to the PET tracer. No serious adverse reactions to this tracer have been reported. Patients may experience some discomfort from having a needle inserted into their arm/hand in order to have the tracer injected. Occasionally the vein may become inflamed or infected, or they may experience bruising at the insertion site. All efforts will be made to avoid or minimise any discomfort or other adverse effects from these procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Age over 18 (no upper limit).
3. Not pregnant.
4. Not breastfeeding.
5. Indeterminate breast lesion on MRI requiring a second-look ultrasound.
6. Ability to lie still for up to 30 minutes prone and supine.
7. Females of childbearing potential have a negative pregnancy test within 7 days prior to being registered. Participants are considered not of child bearing potential if they are surgically sterile (i.e. they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.
8. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Females who are pregnant, planning pregnancy or breastfeeding
2. Concurrent and/or recent involvement in other research that is likely to interfere with the intervention within 3 months prior to study enrolment
3. Inability to lie flat or undergo the tests.
4. Any co-morbidities or conditions which in the opinion of the clinical team means that the patient should be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female only.
Enrollment: 12 (Actual)
Dates: Start 2016-10-05 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-03-04 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Two years.
  To assess the feasibility and acceptability to patients of F-18 FDG breast PET scans, by determining how many patients can be recruited over two years.

SECONDARY OUTCOMES:
Comparison with standard-of-care assessments | Two weeks
  To compare results of breast PET to ultrasound, breast MRI and pathology
Eligibility barriers to recruitment | Two years.
  To determine which eligibility criteria are barriers to recruitment of patients to a study of F-18 FDG breast PET scans.
Comparison with whole-body PET | Two weeks
  To compare the results obtained from F-18 FDG PET CT and breast PET scans
Sample size calculation | Two years.
  To estimate outcome standard deviations to inform sample size calculations for a definitive trial.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wagner, Principal Investigator — Royal Free Hospital NHS Foundation Trust
Locations (1):
- Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All requests for data sharing will adhere to the UCL Surgical & Interventional Trials Unit (SITU) data sharing agreement policy. UCL Medical School is supportive of data sharing and will endeavour to assist in requests for data sharing. These data will be held on secure servers and will not be released to any third parties until all the main outputs from the studies have been published. All requests for access to the data will be formally requested through the use of a SITU data request form which will state the purpose, analysis and publication plans together with the named collaborators. All requests are dealt with on a case by case basis by SITU and the Chief Investigator. All requests will be logged and those successful will have a data transfer agreement which will specify appropriate acknowledgement of the Chief Investigator and study group, the sponsor, and funders.